CLINICAL TRIAL: NCT04258891
Title: Development and Validation of a Multidimensional System to Dynamically Predict Graft Survival After Kidney Transplantation
Brief Title: Multidimensional System to Dynamically Predict Graft Survival After Kidney Transplantation
Acronym: DYNAKT
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: DYNAKT
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Kidney Transplant Failure
Keywords: Kidney Transplantation; Graft survival; Kidney function; Prediction; Dynamic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Kidney recipients aged over 18 and of all sexes recruited from 2004 in European, North American and South American centers, who have estimated glomerular filtration rate and proteinuria follow-up and data from protocol and for cause biopsies for allograft survival assessment; Randomized controlled trials conducted over the past 20 years with available data on protocol biopsy within the first year and follow-up, clinical, biological and histological data.

SUMMARY:
The incidence of end stage renal disease (ESRD) is rapidly increasing, now affecting an estimated 7.4 million people worldwide. Numerous parameters such as demographic, clinical and functional factors drive the deterioration of the kidney, ultimately leading to ESRD. Although some ESRD prediction models have been derived in the past years, none of these models are dynamic: they do not integrate the repeated measurements recorded throughout individuals' follow-up.

As highlighted in several studies, kidney function repeated measurements (i.e., trajectories) are highly associated with graft survival after kidney transplantation. The investigators made the hypothesis that these trajectories may bring relevant information in the context of graft survival risk prediction model. Hence, combining these trajectories with standard graft survival risk factors may enhance prediction performance. This could permit to derive a robust tool that could be updated over time by continuously capturing patient' personal evolution.

DETAILED DESCRIPTION:
850 million individuals suffer from chronic kidney disease (CKD), while diabetes, cancer, and HIV/AIDS affect 422, 42, and 37 million individuals, respectively. End stage renal disease (ESRD) hence places a heavy burden on health systems worldwide. Linked to that, the kidney-disease-associated mortality rate worldwide has risen over the past decade, now causing the death of 5 to 10 million individuals every year.

In kidney transplantation, numerous parameters such as demographic, clinical and functional factors drive the deterioration of the kidney, sometimes leading to graft failure. Current approaches for investigating the relationship between these factors and graft failure have been limited by standard statistical approaches and by registries with an overall lack on granular data, including infrequent kidney function measurements for a single patient and convenience clinical samples. Identifying the determinants of graft failure with a dynamic approach may bring an original perspective to the traditional graft survival risk prediction model that are impeded by their reliance on low-granularity datasets, cross-sectional parameters, and limited follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipients transplanted after 2004
* Kidney recipients over 18 years of age
* Kidney recipients with at least two estimated glomerular filtration rate and proteinuria measurements after transplantation

Exclusion Criteria:

* Combined transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney recipients aged over 18 and of all sexes recruited from 2004 in European and North American centers, who have estimated glomerular filtration rate and proteinuria repeated measurements, data from protocol and for cause biopsies, as well as immunological, clinical, functional parameters and survival data for allograft and patient survival assessment. Additional kidney recipients from RCTs with longitudinal data including baseline and follow-up clinical, functional, immunological and histological data.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Allograft survival probability | Up to 10 years after kidney transplantation
  Allograft survival probability, calculated from a dynamic prediction system, based on clinical, histological, immunological and estimated glomerular filtration rate and proteinuria repeated measurements, assessed at the time of risk evaluation and that can be updated thereafter.

SECONDARY OUTCOMES:
Added prognostic value | Up to 10 years after kidney transplantation
  Added prognostic value of the dynamic prediction system over standard of care monitoring of kidney transplant recipients based on single value of estimated glomerular filtration rate and proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Professor, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (18):
- United States (5):
  - Department of Medicine, Division of Nephrology, Comprehensive Transplant Center, Cedars Sinai Medical Center, Los Angeles, California
  - Division of Transplantation, Department of Surgery, Feinberg School of Medicine, Northwestern University, Chicago, Illinois
  - Department of Surgery, Johns Hopkins University School of Medicine, Baltimore, Maryland
  - William J. von Liebig Center for Transplantation and Clinical Regeneration, Mayo Clinic, Rochester, Minnesota
  - Albert Einstein College of Medicine, Renal Division Montefiore Medical Center, Kidney Transplantation Program, New York, New York
- Unidad de Trasplante Renopáncreas, Centro de Educación Médica e Investigaciones Clínicas, Buenos Aires, Argentina
- Brazil (2):
  - Universidade Federal de São Paulo, Hospital do Rim, Escola Paulista de Medicina, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, Renal Transplantation Service, São Paulo
- Clinica Alemana de Santiago, Santiago, Chile
- Department of Nephrology, Arterial Hypertension, Dialysis and Transplantation, University Hospital Centre Zagreb, School od Medicine University of Zagreb, Zagreb, Croatia
- France (7):
  - Department of Nephrology, Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Nephrology Dialysis Transplantation Department, University of Lorraine, Centre Hospitalier Universitaire de Nancy, Nancy
  - Kidney Transplant Department, Saint-Louis Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Kidney Transplant Department, Necker Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Department of Transplantation, Nephrology and Clinical Immunology, Hôpital Foch, Suresnes
  - Department of Nephrology and Organ Transplantation, Centre Hospitalier Universitaire Rangueil, Toulouse
  - Bretonneau Hospital, Nephrology and Immunology Department, Tours
- Department of Nephrology, Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raynaud M, Aubert O, Divard G, Reese PP, Kamar N, Yoo D, Chin CS, Bailly E, Buchler M, Ladriere M, Le Quintrec M, Delahousse M, Juric I, Basic-Jukic N, Crespo M, Silva HT Jr, Linhares K, Ribeiro de Castro MC, Soler Pujol G, Empana JP, Ulloa C, Akalin E, Bohmig G, Huang E, Stegall MD, Bentall AJ, Montgomery RA, Jordan SC, Oberbauer R, Segev DL, Friedewald JJ, Jouven X, Legendre C, Lefaucheur C, Loupy A. Dynamic prediction of renal survival among deeply phenotyped kidney transplant recipients using artificial intelligence: an observational, international, multicohort study. Lancet Digit Health. 2021 Dec;3(12):e795-e805. doi: 10.1016/S2589-7500(21)00209-0. Epub 2021 Oct 28. PMID 34756569
- See also: Paris Transplant Group Website — https://www.paristransplantgroup.org